CLINICAL TRIAL: NCT01457833
Title: Endoscopic Lung Volume Reduction by Implantation of Endobronchial Valves (EBV) vs. Intrabronchial Valves (IBV) in Patients With Severe Heterogeneous Emphysema
Brief Title: Implantation of Endobronchial Valves Versus Intrabronchial Valves in Patients With Severe Heterogeneous Emphysema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Professor MD, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protokoll E1.0-23.05.2011
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema

ARMS (2):
- Endobronchial valves (EBV) (Active Comparator): Complete occlusion of one emphysematous destroyed lobe by implantation of endobronchial valves
  Interventions: Device: EBV implantation
- Intrabronchial valves (IBV) (Active Comparator): Complete occlusion of one emphysematous destroyed lobe by implantation of intrabronchial valves
  Interventions: Device: IBV implantation

INTERVENTIONS:
Device: EBV implantation — In severe cases of COPD even optimum treatment involving bronchodilatation with drugs, physical training and possibly oxygen therapy is unable to influence exercise capacity and the perception of dyspnoea to a sufficient extent. Given the assumption that the elastic recoil of the small airways can be improved by a reduction in lung volume and pulmonary function overall by more ergonomic breathing mechanics and diaphragm function, various endoscopic procedures for lung volume reduction are available. The most advanced technique is the implantation of valves. The one-way mechanism of these valves allows air to be expelled during exspiration without any influx of air during inspiration.
  Other Names: (Zephyr EBV)
  Arms: Endobronchial valves (EBV)
Device: IBV implantation — In severe cases of COPD even optimum treatment involving bronchodilatation with drugs, physical training and possibly oxygen therapy is unable to influence exercise capacity and the perception of dyspnoea to a sufficient extent. Given the assumption that the elastic recoil of the small airways can be improved by a reduction in lung volume and pulmonary function overall by more ergonomic breathing mechanics and diaphragm function, various endoscopic procedures for lung volume reduction are available. The most advanced technique is the implantation of valves. The one-way mechanism of these valves allows air to be expelled during exspiration without any influx of air during inspiration.
  Other Names: (Spiration IBV)
  Arms: Intrabronchial valves (IBV)

SUMMARY:
Patients with advanced heterogeneous emphysema experience improvement in clinical outcomes in the same way following either implantation of endobronchial valves or intrabronchial valves.

DETAILED DESCRIPTION:
Patient enrollment and data acquisition is to be carried out on a prospective basis. It is planned to enroll a total of 50 patients with advanced heterogeneous emphysema. After decision to undertake endoscopic lung volume reduction by valve implantation patients will be randomised to two treatment arms. 25 patients receive unilateral IBV treatment or unilateral EBV treatment in each case. All patients will undergo treatment at one study centre in Heidelberg.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary function: FEV1 < 45 %, RV > 150 %, TLC > 100 %
* heterogeneous emphysema

Exclusion Criteria:

* homogeneous emphysema
* significant bronchiectasis
* severe concomitant diseases
* pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

PRIMARY OUTCOMES:
Improvement in pulmonary function (FEV1 and RV/TLC) | 6 months

SECONDARY OUTCOMES:
Number of severe adverse events | 6 months
Evaluation of valve migration rate | 6 months
Average changes in pulmonary function (FEV1, IVC, RV, TLC, RV/TLC) | 6 months
Average changes in 6-minute-walk-distance | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany